CLINICAL TRIAL: NCT03429699
Title: Effectiveness of a Stage-based Lifestyle Modification Intervention for Obese Children
Brief Title: Lifestyle Modification Intervention for Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Nor Baizura Md. Yusop, Senior Lecturer, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UPM/FPSK/PADS/T7-MJKEtikalPer
Record Dates: First submitted 2018-02-04; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Childhood Obesity; Life Style Modification
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Stage-based Lifestyle Modification Intervention for the Management of Childhood Obesity
- Control group (Other)
  Interventions: Behavioral: Existing practice for the management of childhood obesity

INTERVENTIONS:
Behavioral: Stage-based Lifestyle Modification Intervention for the Management of Childhood Obesity — The participants will receive treatment based on nutrition clinical practice guideline for the management of childhood obesity. Participants in IG will be received a nutrition clinical practice guideline for the management of childhood obesity that comprised several activities, including nutrition counselling, aerobic sessions, a hands-on activity (healthy food preparation) and 'Sharing is Caring'. The Nutrition Practice Guideline for the Management of Childhood Obesity that comprised recommendations for assessment of nutritional status, determination of energy requirement, dietary prescriptions and physical activity modifications will be used. Participants' SOC for dietary and physical activity behaviors will be determined before any information was given to ensure that the selected educational topic will be tailored to the participant's current SOC.
  Arms: Intervention group
Behavioral: Existing practice for the management of childhood obesity — The participants will receive treatment based on the existing practice for the management of childhood obesity. Only nutritional counseling will be received by CG and standard treatment based on current practices by most dietitians in Malaysia for weight management of obese children will be used.
  Arms: Control group

SUMMARY:
Interventions that encompass behavioral modifications of dietary intake and physical activity dietary management are essential for the management of obese children. This study assessed the effectiveness of a stage-based lifestyle modification intervention for obese children. A total of 50 obese children (7-11 years) were randomized to intervention (n=25) or control (n=25) group. Data were collected at baseline, at follow-up (every month) and at six-month post-intervention. The intervention group (IG) received stage-based lifestyle modification intervention based on Nutrition Practice Guideline for the Management of Childhood Obesity, while the control group (CG) received standard treatment. Changes in body composition, physical activity, and dietary intake were examined in both intervention and control groups.

DETAILED DESCRIPTION:
Main Objective:

To evaluate the effectiveness of Stage-based Lifestyle Modification Intervention for the Management of Childhood Obesity

Specific objectives:

To compare changes in body composition, energy and nutrient intake, as well as physical activity between children receiving the Stage-based Lifestyle Modification Intervention (i.e. intervention group) and the standard treatment (i.e. control group) for the management of childhood obesity.

Study hypothesis:

There is significant different in body mass index (BMI) and body composition, energy and nutrient intakes and physical activity between children receiving nutrition clinical practice guideline (treatment group) and existing management of childhood obesity (control group)?

Interventions Eighty two children will be assigned to two groups, namely Group A (intervention) and Group B (control).

Intervention Group (IG):

The participants will receive treatment based on nutrition clinical practice guideline for the management of childhood obesity. Participants in IG will be received a nutrition clinical practice guideline for the management of childhood obesity that comprised several activities, including nutrition counselling, aerobic sessions, a hands-on activity (healthy food preparation) and 'Sharing is Caring'. The Nutrition Practice Guideline for the Management of Childhood Obesity that comprised recommendations for assessment of nutritional status, determination of energy requirement, dietary prescriptions and physical activity modifications will be used. Participants' SOC for dietary and physical activity behaviours will be determined before any information was given to ensure that the selected educational topic will be tailored to the participant's current SOC. Several educational tools that match participant's current SOC will be used. Nutritional counselling lasted for one hour, and at least two goals for dietary and physical activity will be determined at the end of the session. The researcher (Nor Baizura, M.Y), a trained dietitian, provided nutrition counselling to parents/caregivers and children. An aerobic session will be conducted to encourage participants to be more active and increase their motivation levels, while a hands-on activity is aimed at increasing the knowledge of participants about healthy food preparation. 'Sharing is Caring' session is to encourage parents/caregivers to share their experiences during the intervention period.

b. Control group (CG):

The respondents will receive treatment based on the existing practice for the management of childhood obesity. Only nutritional counselling will be received by CG and standard treatment based on current practices by most dietitians in Malaysia for weight management of obese children will be used. Nutrition counseling is provided by dietitians but not delivered based on SOC as the IG. During nutrition counseling, participants will be assessed and informed about their nutritional status, and this will be followed by advice on dietary intake and physical activity. Participants will be advised to reduce intakes of fats and sweetened drinks, increase intakes of fruits and vegetables, increase physical activity and reduce sedentary activity, but they will not informed specifically about the amounts or quantities of the food to be taken. The nutritional counseling will be conducted for half an hour, and only a related brochure on childhood obesity will be disseminated.

Primary outcome measures: BMI-for-age z-scores Secondary outcome measures: Body composition (waist circumference, mid-upper arm circumference and body fat percentage) - Energy and nutrient intakes (macronutrients, sugar and fiber) -Physical activity

ELIGIBILITY:
Inclusion Criteria:

The participants will be included if they are:

* Children aged 2 - 12 years old
* Obese based on the WHO growth chart 2007 (BMI-for-age more than +2SD)

Exclusion Criteria:

The participants will be excluded if they are:

* Diagnosed with diabetes mellitus, psychiatric disorder (e.g. schizophrenia, severe autism or
* mental retardation or psychosis), or other serious medical conditions.
* Receiving medications that would potentially promote weight gain or weight loss.
* Involved in any weight management program
* Overweight, normal weight and underweight

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-02-02 (Actual); Primary Completion 2014-03-10 (Actual); Study Completion 2014-03-10 (Actual)

PRIMARY OUTCOMES:
weight (kg) | 24 weeks
Height (cm) | 24 weeks
BMI-for-age Z score | 24 weeks

SECONDARY OUTCOMES:
waist circumference (cm) | 24 weeks
Mid-upper Arm Muscle Circumference (cm) | 24 weeks
Body fat (%) | 24 weeks
Energy (kcal) | 24 weeks
carbohydrate (g) | 24 weeks
Protein (g) | 24 weeks
Fat (g) | 24 weeks
Sugar (g) | 24 weeks
Fiber (g) | 24 weeks
Physical Activity Questionnaire for Older Children (PAQ-C) | 24 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Md Yusop NB, Mohd Shariff Z, Hwu TT, Abd Talib R, Spurrier N. The effectiveness of a stage-based lifestyle modification intervention for obese children. BMC Public Health. 2018 Mar 1;18(1):299. doi: 10.1186/s12889-018-5206-2. PMID 29490648